CLINICAL TRIAL: NCT04238273
Title: Hemodynamic Changes With Heated, Humidified High Flow Nasal Cannula (HHHFNC) Versus Nasal Continuous Positive Airway Pressure (nCPAP) for Respiratory Support of Preterm Neonates
Brief Title: High Flow Nasal Cannula Versus Nasal Continuous Positive Airway Pressure for Respiratory Support of Preterm Neonates
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, Professor, Ain Shams University
Other Study IDs: FMASU MD 386/2017
Record Dates: First submitted 2020-01-09; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Hemodynamic changes; High flow nasal cannula; Nasal continuous positive airway pressure; Respiratory distress syndrome; Prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HHHFNC: it included 63 preterm neonates on Heated, Humidified High Flow Nasal Cannula, of which 35 preterm underwent functional echocardiography, transcranial ultrasonography Doppler applied to the anterior cerebral artery and assessment of pre-prandial superior mesenteric artery velocity and volume of blood flow with Doppler sonography. All of which done while on non invasive ventilation and after weaning.
  Interventions: Diagnostic Test: Functional Echocardiography
- NCPAP: it included 60 preterm neonates on Nasal Continuous Positive Airway Pressure, of which 35 preterm underwent functional echocardiography, transcranial ultrasonography Doppler applied to the anterior cerebral artery and assessment of pre-prandial superior mesenteric artery velocity and volume of blood flow with Doppler sonography. All of which done while on non invasive ventilation and after weaning.
  Interventions: Diagnostic Test: Functional Echocardiography

INTERVENTIONS:
Diagnostic Test: Functional Echocardiography — Imaging studies to assess Hemodynamics of both groups on and off non invasive ventilation
  Other Names: Transcranial ultrasonography Doppler applied to the anterior cerebral artery; Assessment of pre-prandial superior mesenteric artery velocity and volume of blood flow with Doppler sonography

SUMMARY:
This work is designed to:

1. Evaluate the efficacy of HHHFNC in comparison with nCPAP in preterm neonates.
2. Investigate hemodynamic changes associated with HHHFNC in comparison to nCPAP in preterm neonates during periods of non-invasive respiratory support and after being off support.

DETAILED DESCRIPTION:
There is a preference of using noninvasive modes of ventilation for management of respiratory distress syndrome (RDS) in preterm infants and of weaning of ventilated neonates as soon as possible to non-invasive modes.

Yet, little is known about which non-invasive mode is better and the hemodynamic changes that occur to the infants secondary to these modes. The study provides an evaluation of the efficacy of heated, humidified high flow nasal cannula (HHHFNC) in comparison to nasal continuous positive airway pressure (nCPAP) in preterm infants. Secondary aim is to assess echographic, cerebral blood flow and mesenteric blood flow changes during HHHFNC versus nCPAP.

ELIGIBILITY:
Inclusion Criteria:

Infants are eligible if they meet the following criteria:

1. Gestational age ≤ 35 weeks.
2. Preterm neonates in need for non invasive ventilation whether they were on invasive ventilatory support before or not.

Exclusion Criteria:

Preterm neonates with evidence of any of the following will be excluded:

1. Major upper or lower airway anomalies.
2. Significant congenital anomalies including cardiac, abdominal or respiratory.
3. Hemodynamically significant patent ductus arteriosus (PDA): diagnosed if there is colour doppler echocardiographic evidence of left to right ductal shunt, ductal diameter >1.5mm/kg or left atrial/aortic root ratio >1.4

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted on preterm neonates who required ventilatory support for respiratory distress syndrome (RDS) with previous invasive ventilation or not. The involved study group will be of matched gestational, postnatal age and sex.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Echocardiography study for preterm neonates among the two study groups while on and off non invasive ventilation. | 2 years
  Done using Bedside functional echocardiography to record Superior vena caval flow (ml/kg/min), right ventricular output flow (ml/kg/min) and left ventricular output flow (ml/kg/min) for each preterm neonate in one of the two study groups (using either HHHFNC and nCPAP) on and off respiratory support.

SECONDARY OUTCOMES:
Evaluate the efficacy of HHHFNC in comparison with nCPAP in preterm neonates. | 2 years
  The percentage of success and failure among the HHHFNC and nCPAP groups , success defined as the preterm neonate that will not require invasive ventilation, while failure as the preterm neonate that will require invasive ventilation.
Anterior cerebral artery Doppler (measuring resistive index) and preprandial Superior mesenteric artery Doppler (measuring resistive index). | 2 years
  Anterior cerebral artery resistive index and preprandial Superior mesenteric artery resistive index measured for 70 preterm neonate on and off non invasive ventilation. 35 preterm placed on HHHFNC in comparison to 35 preterm placed on nCPAP.
Preprandial Superior mesenteric artery Doppler measuring superior mesenteric artery blood flow(mL/sec) | 2 years
  Preprandial Superior mesenteric artery blood flow(mL/sec) measured for 70 preterm neonate on and off non invasive ventilation. 35 preterm placed on HHHFNC in comparison to 35 preterm placed on nCPAP.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Hisham Abdel Samie Awad, Study Director — Ain Shams University,Medical school, Pediatrics department
Locations (1):
- 38 abbasia, next to nour mosque, Ain Shams University Hospital, Pediatrics department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided